CLINICAL TRIAL: NCT03964454
Title: Individual Breastfeeding Support With Contingent Incentives for Low-Income Mothers
Brief Title: BOOST: Breastfeeding Onset and Onward With Support Tools
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Temple University (Other); Christiana Care Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BOOST; R01HD094877 (NIH)
Record Dates: First submitted 2019-05-22; First posted 2019-05-28 (Actual); Results first posted 2025-01-01 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Breastfeeding Duration
Keywords: Breastfeeding duration; WIC; low-income; health incentives

STUDY DESIGN:
Intervention Model Description: This is a two-group parallel randomized controlled trial testing the efficacy of health incentives to increase breastfeeding duration among low income WIC eligible mothers.
Who Masked: Outcomes Assessor
Masking Description: Those who are providing home visitations on a monthly basis will be blinded to which condition a participant gets randomized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SC + BFI (Experimental): Participants randomized into SC+BFI will receive the same services as the Standard Care Control (SC) group (standard breastfeeding services from Special Supplemental Nutrition Program for Women, Infants, and Children (WIC) plus monthly home visits that facilitate navigation to as-needed resources and referrals to services that support breastfeeding and problem solving) plus financial incentives contingent on observed breastfeeding.
  Interventions: Behavioral: WIC support + home-based individual support + Breastfeeding Incentives (SC+BFI)
- SC (Active Comparator): Participants randomized into Standard Care (SC) will receive standard breastfeeding services from Special Supplemental Nutrition Program for Women, Infants, and Children (WIC) plus monthly home visits that facilitate navigation to as-needed resources and referrals to services that support breastfeeding and problem solving.
  Interventions: Behavioral: WIC support + home-based individual support (SC)

INTERVENTIONS:
Behavioral: WIC support + home-based individual support + Breastfeeding Incentives (SC+BFI) — Participants randomized into SC+BFI will receive the same services as the Standard Care Control (SC) group (standard breastfeeding services from Special Supplemental Nutrition Program for Women, Infants, and Children (WIC) plus monthly home visits that facilitate navigation to as-needed resources and referrals to services that support breastfeeding and problem solving) plus financial incentives (Breastfeeding Incentives, BFI) contingent on observed breastfeeding.
  Arms: SC + BFI
Behavioral: WIC support + home-based individual support (SC) — Participants randomized into SC will receive standard breastfeeding services from Special Supplemental Nutrition Program for Women, Infants, and Children (WIC) plus monthly home visits that facilitate navigation to as-needed resources and referrals to services that support breastfeeding and problem solving.
  Arms: SC

SUMMARY:
This behavioral intervention trial will test whether a standard care breastfeeding intervention from the Special Supplemental Nutrition Program for Women, Infants, and Children (WIC) program plus monthly financial incentives contingent on observed breastfeeding will improve breastfeeding duration among low-income mothers compared to a standard (WIC) care control. Investigators hypothesize that the standard care plus monthly contingent financial incentives intervention will promote longer breastfeeding duration, fewer infant health issues, and greater healthcare cost savings than the standard care (control) intervention.

DETAILED DESCRIPTION:
Low-income racial/ethnic-minority women have greater challenges with breastfeeding uptake and duration than the general population, resulting in an average breastfeeding duration of four months. This duration is substantially shorter than evidence-based recommendations by the American Academy of Pediatrics to exclusively breastfeed for six months in addition to continued breastfeeding through the first year. Insufficient duration of any breastfeeding is related to multiple maternal and child health problems and increases in breastfeeding duration could be cost saving medically and societally.

Even though breastfeeding counseling and peer support have been effective in prolonging breastfeeding duration in the general maternal population, the effect has not been as strong for WIC-eligible (Special Supplemental Nutrition Program for Women, Infants, and Children (WIC)), low-income mothers. Examining novel adjunctive intervention components that could enhance standard WIC counseling and support is warranted. We tested an incentive-based intervention among low-income Puerto Rican mothers in a pilot study. Results suggested strong potential for efficacy of monthly financial incentives contingent on observed breastfeeding for 6 months combined with WIC usual care, compared to WIC usual care only.

The current, full-scale randomized trial will test the efficacy and generalizability of the 6-month incentive-based approach to increase breastfeeding duration in WIC-eligible mothers through 12 months. The aims of the study are guided by the mission of NICHD's Pregnancy and Perinatology Branch to improve the long-term maternal and infant health of low-income populations via encouraging breastfeeding in the translational research context.

This study is a 2-group, multi-site, parallel randomized controlled trial. The study will be conducted in two regional sites with high concentrations of low-income racial/ethnic minority mothers, Philadelphia, PA and Newark, DE. Participants (n=168) include WIC-eligible mothers who will be allocated into one of the two study groups: (1) A Standard Care Control (SC) group consisting of breastfeeding support through WIC, with home-based individual support, or (2) Standard Care plus Incentives contingent on demonstrating successful breastfeeding (SC+BFI).

Participants randomized into SC will receive standard breastfeeding services from WIC plus monthly home visits that facilitate navigation to as-needed resources and referrals to services that support breastfeeding and problem solving. Participants randomized into SC+BFI will receive the same WIC services and monthly home visits as the SC group, with addition of financial incentives following each home visit that are contingent on observed breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

* mothers must initiate breastfeeding
* mothers must be WIC-enrolled or eligible to enroll in WIC services
* mothers must reside and plan to stay in the study county for 12 months postpartum
* mothers must consent voluntarily
* mothers must understand fifth grade level of English
* mothers must be at least 18 years old

Exclusion Criteria:

* mothers whose babies are medically contraindicated against breastfeeding
* mothers who are hospitalized for severe postpartum medical issues
* mothers who have ongoing illicit drug use issues
* mothers who had a psychiatric hospitalization within the last three months
* mothers who currently have suicidal thoughts or attempts

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 168 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2025-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yukiko Washio, PhD, Principal Investigator — RTI International
Locations (2):
- United States (2):
  - Christiana Care Health Services, Inc., Newark, Delaware
  - Temple University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
A limited data set in which names and other personal health identifiers are removed, as defined by the Health Insurance Portability and Accountability Act (HIPAA), will be supplied to researchers on request.
Time Frame: The data will be made available after the publication of the study results.
Access Criteria: Analytic files will be collected in Redcap and then prepared in SPSS, R, SAS, or STATA, with online codebooks giving the variable name, label, type, format, positions, consistency codes, and, if applicable, values and value labels. Requesting access to data will involve drafting an abstract, checking the feasibility relative to the available data, and then seeking the permission of the PI and the team for review, if appropriate. The data sets will be ready for use and can be converted to other analytic tools.

REFERENCES:
- [Derived] Washio Y, Collins BN, Hunt-Johnson A, Zhang Z, Herrine G, Hoffman M, Kilby L, Chapman D, Furman LM. Individual breastfeeding support with contingent incentives for low-income mothers in the USA: the 'BOOST (Breastfeeding Onset & Onward with Support Tools)' randomised controlled trial protocol. BMJ Open. 2020 Jun 16;10(6):e034510. doi: 10.1136/bmjopen-2019-034510. PMID 32554737

RESULTS

PARTICIPANT FLOW:
Groups:
- WIC Support + Home-based Individual Support + Breastfeeding Incentives (SC+BFI): Participants randomized into SC+BFI will receive the same services as the Standard Care Control (SC) group (standard breastfeeding services from Special Supplemental Nutrition Program for Women, Infants, and Children (WIC) plus monthly home visits that facilitate navigation to as-needed resources and referrals to services that support breastfeeding and problem solving) plus financial incentives contingent on observed breastfeeding.
  WIC support + home-based individual support + Breastfeeding Incentives (SC+BFI): Participants randomized into SC+BFI will receive the same services as the Standard Care Control (SC) group (standard breastfeeding services from Special Supplemental Nutrition Program for Women, Infants, and Children (WIC) plus monthly home visits that facilitate navigation to as-needed resources and referrals to services that support breastfeeding and problem solving) plus financial incentives (Breastfeeding Incentives, BFI) contingent on observed breastfeeding.
- Standard Care as WIC Support + Home-based Individual Support (SC): Participants randomized into Standard Care (SC) will receive standard breastfeeding services from Special Supplemental Nutrition Program for Women, Infants, and Children (WIC) plus monthly home visits that facilitate navigation to as-needed resources and referrals to services that support breastfeeding and problem solving.
  WIC support + home-based individual support (SC): Participants randomized into SC will receive standard breastfeeding services from Special Supplemental Nutrition Program for Women, Infants, and Children (WIC) plus monthly home visits that facilitate navigation to as-needed resources and referrals to services that support breastfeeding and problem solving.
Period: Overall Study
Arm/Group | WIC Support + Home-based Individual Support + Breastfeeding Incentives (SC+BFI) | Standard Care as WIC Support + Home-based Individual Support (SC)
Started | 85 | 83
Completed | 68 | 65
Not Completed | 17 | 18
Not completed — Lost to Follow-up | 13 | 7
Not completed — Withdrawal by Subject | 4 | 11

BASELINE CHARACTERISTICS:
Groups:
- WIC Support + Home-based Individual Support + Breastfeeding Incentives (SC + BFI): Participants randomized into SC+BFI will receive the same services as the Standard Care Control (SC) group (standard breastfeeding services from Special Supplemental Nutrition Program for Women, Infants, and Children (WIC) plus monthly home visits that facilitate navigation to as-needed resources and referrals to services that support breastfeeding and problem solving) plus financial incentives contingent on observed breastfeeding.
  WIC support + home-based individual support + Breastfeeding Incentives (SC+BFI): Participants randomized into SC+BFI will receive the same services as the Standard Care Control (SC) group (standard breastfeeding services from Special Supplemental Nutrition Program for Women, Infants, and Children (WIC) plus monthly home visits that facilitate navigation to as-needed resources and referrals to services that support breastfeeding and problem solving) plus financial incentives (Breastfeeding Incentives, BFI) contingent on observed breastfeeding.
- Total: Total of all reporting groups
Arm/Group | WIC Support + Home-based Individual Support + Breastfeeding Incentives (SC + BFI) | Standard Care as WIC Support + Home-based Individual Support (SC) | Total
Number analyzed (Participants) | 85 | 83 | 168
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.8 (6) | 27.3 (5.1) | 27.6 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 83 | 168
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic White | 6 | 5 | 11
  Hispanic Black | 4 | 4 | 8
  Hispanic Other | 21 | 21 | 42
  Non-Hispanic White | 4 | 1 | 5
  Non-Hispanic Black | 47 | 49 | 96
  Non-Hispanic Other | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 85 | 83 | 168
Relationship status [Count of Participants; unit: Participants]
  Single, never married | 65 | 64 | 129
  Married | 13 | 16 | 29
  Other | 7 | 3 | 10
Years of schooling [Mean (Standard Deviation); unit: years] | 13.1 (2.3) | 13.2 (2.1) | 13.2 (2.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Breastfeeding Their Infants at 1 Month
Description: Identify breastfeeding behavior via standardized observational method: Identifying audible swallowing, regular suck/swallow/breathe pattern, or visible milk in the infant's mouth.
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | WIC Support + Home-based Individual Support + Breastfeeding Incentives (SC+BFI) | Standard Care as WIC Support + Home-based Individual Support (SC)
Number analyzed (Participants) | 81 | 80
Participants | 76 | 74

2. Primary Outcome: Number of Participants Breastfeeding Their Infants at 3 Months
Description: as for outcome 1
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | WIC Support + Home-based Individual Support + Breastfeeding Incentives (SC + BFI) | Standard Care as WIC Support + Home-based Individual Support (SC)
Number analyzed (Participants) | 76 | 75
Participants | 59 | 53

3. Primary Outcome: Number of Participants Breastfeeding Their Infants at 6 Months
Description: as for outcome 1
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | WIC Support + Home-based Individual Support + Breastfeeding Incentives (SC + BFI) | Standard Care as WIC Support + Home-based Individual Support (SC)
Number analyzed (Participants) | 76 | 68
Participants | 46 | 33

4. Primary Outcome: Number of Participants Breastfeeding Their Infants at 9 Months
Description: as for outcome 1
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | WIC Support + Home-based Individual Support + Breastfeeding Incentives (SC + BFI) | Standard Care as WIC Support + Home-based Individual Support (SC)
Number analyzed (Participants) | 69 | 66
Participants | 26 | 19

5. Primary Outcome: Number of Participants Breastfeeding Their Infants at 12 Months
Description: as for outcome 1
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | WIC Support + Home-based Individual Support + Breastfeeding Incentives (SC + BFI) | Standard Care as WIC Support + Home-based Individual Support (SC)
Number analyzed (Participants) | 70 | 65
Participants | 21 | 15

6. Secondary Outcome: Infant Weight
Description: Measured with a portable digital infant scale.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: grams
Groups:
- WIC Support + Home-based Individual Support + Breastfeeding Incentives (SC + BFI): WIC support + home-based individual support + Breastfeeding Incentives (SC+BFI): Participants randomized into SC+BFI will receive the same services as the Standard Care Control (SC) group (standard breastfeeding services from Special Supplemental Nutrition Program for Women, Infants, and Children (WIC) plus monthly home visits that facilitate navigation to as-needed resources and referrals to services that support breastfeeding and problem solving) plus financial incentives (Breastfeeding Incentives, BFI) contingent on observed breastfeeding.
- Standard Care as WIC Support + Home-based Individual Support (SC): WIC support + home-based individual support (SC): Participants randomized into SC will receive standard breastfeeding services from Special Supplemental Nutrition Program for Women, Infants, and Children (WIC) plus monthly home visits that facilitate navigation to as-needed resources and referrals to services that support breastfeeding and problem solving.
Arm/Group | WIC Support + Home-based Individual Support + Breastfeeding Incentives (SC + BFI) | Standard Care as WIC Support + Home-based Individual Support (SC)
Number analyzed (Participants) | 66 | 68
grams | 6199 (1003) | 5921 (886)

7. Secondary Outcome: Infant Weight
Description: Measured with a portable digital infant scale.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | WIC Support + Home-based Individual Support + Breastfeeding Incentives (SC + BFI) | Standard Care as WIC Support + Home-based Individual Support (SC)
Number analyzed (Participants) | 68 | 61
grams | 8099 (1355) | 7943 (1136)

8. Secondary Outcome: Infant Weight
Description: Measured with a portable digital infant scale.
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | WIC Support + Home-based Individual Support + Breastfeeding Incentives (SC + BFI) | Standard Care as WIC Support + Home-based Individual Support (SC)
Number analyzed (Participants) | 67 | 62
grams | 9310 (1591) | 8948 (1151)

9. Secondary Outcome: Infant Weight
Description: Measured with a portable digital infant scale.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | WIC Support + Home-based Individual Support + Breastfeeding Incentives (SC + BFI) | Standard Care as WIC Support + Home-based Individual Support (SC)
Number analyzed (Participants) | 65 | 61
grams | 10101 (1700) | 10018 (1422)

10. Secondary Outcome: Infant Weight
Description: Measured with a portable digital infant scale.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | WIC Support + Home-based Individual Support + Breastfeeding Incentives (SC + BFI) | Standard Care as WIC Support + Home-based Individual Support (SC)
Number analyzed (Participants) | 78 | 75
grams | 4090 (687) | 4241 (711)

ADVERSE EVENTS:
Time Frame: 12 months per participant
Arm/Group | WIC Support + Home-based Individual Support + Breastfeeding Incentives (SC+BFI) | Standard Care as WIC Support + Home-based Individual Support (SC)
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/83
Serious Adverse Events (participants affected / at risk) | 0/85 | 5/83
Other Adverse Events (participants affected / at risk) | 19/85 | 26/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | WIC Support + Home-based Individual Support + Breastfeeding Incentives (SC+BFI) (N=85) | Standard Care as WIC Support + Home-based Individual Support (SC) (N=83)
Hospitailzation of participant (Injury, poisoning and procedural complications) | 0 | 2
Hospitalization of infant (Infections and infestations) | 0 | 2
Infant death (General disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | WIC Support + Home-based Individual Support + Breastfeeding Incentives (SC+BFI) (N=85) | Standard Care as WIC Support + Home-based Individual Support (SC) (N=83)
Depression (Psychiatric disorders) | 6 | 12
Homelessness (Pregnancy, puerperium and perinatal conditions) | 0 | 2
Miscarriage (Pregnancy, puerperium and perinatal conditions) | 1 | 2
COVID infection (Infections and infestations) | 0 | 6
Domestic abuse (Psychiatric disorders) | 3 | 2
ER visit (Infections and infestations) | 2 | 1
Breast cancer or breast issue (Reproductive system and breast disorders) | 1 | 1
Accident (Musculoskeletal and connective tissue disorders) | 1 | 0
Family death or separation (Social circumstances) | 4 | 0
Incarceration (Social circumstances) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-03): https://cdn.clinicaltrials.gov/large-docs/54/NCT03964454/Prot_SAP_000.pdf